CLINICAL TRIAL: NCT03443258
Title: Needs Assessment and Decision-making Tool (NEAT-decision) Integrated in a Clinical Practice to Enhance Patient Involvement in Head and Neck Cancer Rehabilitation - a Randomized Controlled Trial
Brief Title: Needs Assessment Tool Integrated in Clinical Practice of Head and Neck Cancer Rehabilitation
Acronym: NEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Novo Nordisk A/S (Industry); Danish Nurses Organisation (Other)
Responsible Party: Principal Investigator, Annelise Mortensen, PhD student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 05781
Record Dates: First submitted 2018-01-31; First posted 2018-02-23 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients are assigned to either intervention or control group. The intervention group receives a nursing consultation using a need assessment and decision making tool. The control group receives usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (IG) (Experimental): Patients receive needs assessment tool integrated in nursing consultation in accordance with requirements by Danish Health and Medicine Board follow-up program for HNC patients. The consultation consists of 6 steps 1. Welcoming patient; 2. Introducing patient to assessment tool; 3. Discuss symptoms and concerns patient wishes to discuss; 4. Follow up on patients symptoms, concerns and emotional reactions/problems; 5. Accompany/support patient during appointment with surgeon and in cooperation with patient and surgeon ensure that problems arising from the tool needing medical attention are focused on; 6. Continue the consultation after appointment with surgeon; refer patient to multi-disciplinary team members when needed
  Interventions: Other: Needs assesment tool integrated in nursing consultation.
- Control Group (CG) (No Intervention): CG will receive standard care according to the Danish Health and Medicine Board's follow-up program for HNC patients. At present this is done by a staff nurse interviewing the patient, who is a member of the rehabilitation team who perform nursing consultations. The interview takes place after the appointment with the surgeon. The nurse refers the patient to physical rehabilitation if needed

INTERVENTIONS:
Other: Needs assesment tool integrated in nursing consultation. — Needs assessment tool consisting of 57 items related to functional, emotional, social and existential areas guide follow-up care and referral to multidisciplinary team rehabilitation e.g. dietician; speech-pathologist; psychologist, etc
  Arms: Intervention Group (IG)

SUMMARY:
The study tests a needs assessment and decision-making tool with patients who are in need of rehabilitation after surgery for Head and Neck Cancer. The purpose is to enhance patient involvement in decision-making.

DETAILED DESCRIPTION:
The study tests a needs assessment and decision-making tool with patients surgically treated for Head and Neck Cancer. The tool will be an integrated part of a new clinical practice with nursing consultations at three seperate time-points in the post-surgical period of the patients. Half of the participants will receive nursing consultations using the tool and the other half will receive standard care.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Head and Neck Cancer
* Stage T3 or T4
* Surgically treated
* Must be able to speak and understand Danish

Exclusion Criteria:

* Treated surgically for thyroid or parotic cancers
* Referred to adjuvant radio - or chemotherapy
* Having an unstable psychiatric illness.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Health Related Quality of Life, from baseline to 9, 21 and until 67 days post surgery | Baseline; 9; 21 and 67 days post-surgery
  Questionnaire measuring 35 items related to quality of life in head and neck cancer. European Organisation for Research and Treatment of Cancer Quality of Life and Head and Neck Cancer (EORTC QLQ-H&N35). Scores range from 0 - 100,, where a high score represents high quality of life. The study will measure global quality of life

SECONDARY OUTCOMES:
Change in Symptom Burden from baseline to 2, 14 and 60 days post-surgery | Baseline, 2, 14 and 60 days post-surgery
  Questionnaire measuiring 28 items related to symptoms of head and neck cancer patients. MD Anderson Symptom Inventory Head and Neck Cancer module (MDASI-HN). Scores range from 0 - 10, where a high score represents a high symptom burden interference with daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Annelise Mortensen, MSA, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Dept. Of Otorhinolaryngology, Head and Neck Surgery and Audiology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mortensen A, Wessel I, Rogers SN, Tolver A, Jarden M. Needs assessment in patients surgically treated for head and neck cancer-a randomized controlled trial. Support Care Cancer. 2022 May;30(5):4201-4218. doi: 10.1007/s00520-021-06759-9. Epub 2022 Jan 27. PMID 35083545

DOCUMENTS (1):
  • Study Protocol (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT03443258/Prot_000.pdf